CLINICAL TRIAL: NCT05956158
Title: RISE: A Remote Study of Insomnia Treatment in Crohn's Disease
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jessica.K.Salwen-Deremer, Assistant Professor of Psychiatry & Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY02001855
Record Dates: First submitted 2023-06-22; First posted 2023-07-21 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Insomnia; Crohn Disease
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Crohn Disease | interventions — Behavior Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Treatment (Experimental)
  Interventions: Behavioral: Behavioral Treatment
- Sleep Education Treatment (Placebo Comparator)
  Interventions: Behavioral: Sleep Education Treatment

INTERVENTIONS:
Behavioral: Behavioral Treatment — This treatment is designed to help participants make changes to behavior patterns and thoughts that contribute to insomnia.
  Other Names: Cognitive Behavioral Therapy for Insomnia; CBT-I
  Arms: Behavioral Treatment
Behavioral: Sleep Education Treatment — This treatment is designed to help participants understand the relationships among sleep, pain, and Crohn's disease and to make changes to insomnia-related behaviors.
  Arms: Sleep Education Treatment

SUMMARY:
The purpose of this study is to assess whether the investigators can treat insomnia in people with Crohn's disease, and if insomnia treatment can make other things better, like pain or inflammation.

DETAILED DESCRIPTION:
People with Crohn's disease often suffer from sleep problems. Long term, sleep problems may lead to more flares of Crohn's disease or other complications. In general, patients with Crohn's disease also report that sleep problems can worsen symptoms of Crohn's disease the next day. In people with other medical problems, research has also shown that having sleep problems can make other things worse, such as pain and inflammation. In this study, the investigators want to understand if they can treat sleep problems in people with Crohn's disease, and what else might improve if sleep gets better. If this study is successful, it will help the investigators understand more about how to treat insomnia in people with Crohn's disease and how sleep impacts pain and inflammation. Long term, this information will be helpful in understanding how best to take care of people with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate CD based on PRO-3 & 50% with objective evidence of active disease
* Insomnia Severity Index score ≥ 8 and SOL or WASO ≥ 30 minutes
* Stability of sleep & CD meds for ≥ 3 months
* Access to internet or cell phone service sufficient for telehealth

Exclusion Criteria:

* PHQ-9 depression score ≥ 15
* GAD-7 anxiety score ≥ 15
* Unstable major psychiatric condition (e.g., bipolar disorder, psychotic disorder)
* Current alcohol or substance abuse
* Current opioid use for pain control
* Current systemic corticosteroid use
* Current pregnancy or nursing
* Ileostomy or colostomy
* Diagnosis of seizure disorder
* Diagnosis of sleep apnea or positive WatchPAT screen
* Diagnosis of restless leg syndrome or positive Cambridge-Hopkins RSLq screen
* Night shift, rotating shift work, or frequent travel outside of time zone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention as measured by attrition rate over time | Baseline, 8 weeks, 21 weeks, and 34 weeks
  Attrition rate will be based on the percentage of participants who have dropped out of the trial at different time points.
Feasibility of the intervention as measured by recruitment rate over time | From study initiation until we are no longer actively recruiting (approximately 24 months)
  Recruitment rate will be based on the number of participants who are recruited into the trial per month.
Feasibility of the intervention as measured by assessment completion at multiple time points | Baseline, 8 weeks, 21 weeks, and 34 weeks
  Assessment completion rate will be based on the percentage of participants who complete all the required questionnaires and tasks at each time point.
Feasibility of the intervention as measured by qualitative interviews | 8 weeks and 34 weeks
  Feasibility will be based on interview-derived themes related to barriers and facilitators to study engagement. Data will be collected at two time points to ensure completeness of themes.
Acceptability of the intervention as measured by visit completion | 8 weeks
  Visit completion will be based the number of visits (out of 5) completed by each participant.
Treatment acceptability questionnaire score | 1 week
  The Treatment Acceptability Questionnaire is a 4-item self-report questionnaire designed to assess the overall acceptability of an intervention. Scores range from 1 to 4 and higher scores are indicative of greater acceptability.
Acceptability of the intervention as measured by qualitative interviews | 8 weeks
  Acceptability will be based on interview-derived themes related to aspects of the intervention that participants found helpful and unhelpful.

SECONDARY OUTCOMES:
Change in insomnia symptoms as measured by the Insomnia Severity Index | Baseline, 8 weeks, 21 weeks, and 34 weeks
  The Insomnia Severity Index (ISI) is a self-report questionnaire designed to measure severity of insomnia. The ISI is made up of 7 items on insomnia symptoms and related impairments and total scores range from 0-28. Higher scores are indicative of greater insomnia symptoms.
Change in diary-based sleep onset latency | Baseline, 8 weeks, 21 weeks, and 34 weeks
  A weekly average of self-reported time it takes to fall asleep each night, derived from a self-reported sleep diary
Change in diary-based wake after sleep onset | Baseline, 8 weeks, 21 weeks, and 34 weeks
  A weekly average of self-reported time spent awake in the middle of each night, derived from a self-reported sleep diary
Change in Crohn's disease symptoms as measured by the Patient Reported Outcomes 3 | Baseline, 8 weeks, 21 weeks, and 34 weeks
  The Patient Reported Outcomes 3 (PRO-3) is a self-report questionnaire designed to measure the severity of Crohn's disease symptoms in the past week. The PRO-3 is made up of 3 items (stool frequency, pain, and well-being) and higher scores are indicative of more severe symptoms. Scores are interpreted as follows: <13=quiescent or inactive disease; 13-21=mildly active disease; 22-52=moderately active disease; 53 and up=severely active disease.

OTHER OUTCOMES:
Change in C-reactive protein | Baseline, 8 weeks, and 21 weeks
  We will measure blood levels of C-reactive protein
Change in fecal calprotectin | Baseline, 8 weeks, and 21 weeks
  We will measure levels of fecal calprotectin via a stool sample.
Change in sleep architecture | Baseline, 8 weeks, and 21 weeks
  We will measure changes in percent time spent in light sleep, deep sleep, and rapid eye movement (REM) sleep using the Oura ring.
Change in behaviorally assessed pain tolerance via the Cold Pressor Test | Baseline, 8 weeks, and 21 weeks
  The Cold Pressor Test involves submerging one's non-dominant hand in ice water and rating discomfort at regular, pre-determined intervals. Pain tolerance will be measured based on the total amount of time a participant can keep their hand submerged, with a maximum of 3 minutes.
Change in diary-based sleep efficiency | Baseline, 8 weeks, 21 weeks, and 34 weeks
  Change in sleep efficiency (total sleep time / time in bed), derived from a self-reported sleep diary.
Change in objective sleep onset latency | Baseline, 8 weeks, and 21 weeks
  Change in the time it takes to fall asleep each night, derived from the Oura ring.
Change in objective wake after sleep onset | Baseline, 8 weeks, and 21 weeks
  Change in the time spent awake in the middle of the night, derived from the Oura ring.
Change in objective sleep efficiency | Baseline, 8 weeks, and 21 weeks
  Change in sleep efficiency (total sleep time / time in bed), derived from the Oura ring.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided